CLINICAL TRIAL: NCT02900859
Title: Infraorbital Nerve Involvement on Magnetic Resonance Imaging in European Patients With IgG4-related Ophthalmic Disease
Acronym: RetroG4
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: NI_ALR_2015_2
Record Dates: First submitted 2016-09-06; First posted 2016-09-14 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Orbital Inflammation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

SUMMARY:
Systematic medical chart and imaging files review of patients presenting with non-lymphoma, non-thyroid-related orbital inflammation. The review aims at comparing the frequency of MRI infra-orbital nerve enlargement, between patients diagnosed with an IgG4-related ophthalmic disease (IgG4-ROD) and other patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient suffering from acute orbital inflammation

Exclusion Criteria:

* Thyroid disease
* Lymphoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from non-lymphoma, non-thyroid-related orbital inflammation
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2006-01; Primary Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Infra-orbital nerve enlargement on orbital MRI | Within 1 week following diagnosis